CLINICAL TRIAL: NCT04313647
Title: A Tolerance Clinical Study On Aerosol Inhalation of Mesenchymal Stem Cells Exosomes In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEXVT
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Results first posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: mesenchymal stem cells; exosomes; mesh nebulizer

STUDY DESIGN:
Intervention Model Description: MSCs-exosomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1X level (Experimental): Aerosol inhalation of MSCs-derived exosomes treatment participants will receive once aerosol inhalation of MSCs-derived exosomes (2.0*10^8 nano vesicles/3 ml)
  Interventions: Biological: 1X level of MSCs-Exo
- 2X level (Experimental): Aerosol inhalation of MSCs-derived exosomes treatment participants will receive once aerosol inhalation of MSCs-derived exosomes (4.0*10^8 nano vesicles/3 ml)
  Interventions: Biological: 2X level of MSCs-Exo
- 4X level (Experimental): Aerosol inhalation of MSCs-derived exosomes treatment participants will receive once aerosol inhalation of MSCs-derived exosomes (8.0*10^8 nano vesicles/3 ml)
  Interventions: Biological: 4X level of MSCs-Exo
- 6X level (Experimental): Aerosol inhalation of MSCs-derived exosomes treatment participants will receive once aerosol inhalation of MSCs-derived exosomes (12.0*10^8 nano vesicles/3 ml)
  Interventions: Biological: 6X level of MSCs-Exo
- 8X level (Experimental): Aerosol inhalation of MSCs-derived exosomes treatment participants will receive once aerosol inhalation of MSCs-derived exosomes (16.0*10^8 nano vesicles/3 ml)
  Interventions: Biological: 8X level of MSCs-Exo

INTERVENTIONS:
Biological: 1X level of MSCs-Exo — Once aerosol inhalation of MSCs-derived exosomes (2.0*10^8 nano vesicles/3 ml)
  Arms: 1X level
Biological: 2X level of MSCs-Exo — Once aerosol inhalation of MSCs-derived exosomes (4.0*10^8 nano vesicles/3 ml)
  Arms: 2X level
Biological: 4X level of MSCs-Exo — Once aerosol inhalation of MSCs-derived exosomes (8.0*10^8 nano vesicles/3 ml)
  Arms: 4X level
Biological: 6X level of MSCs-Exo — Once aerosol inhalation of MSCs-derived exosomes (12.0*10^8 nano vesicles/3 ml)
  Arms: 6X level
Biological: 8X level of MSCs-Exo — Once aerosol inhalation of MSCs-derived exosomes (16.0*10^8 nano vesicles/3 ml)
  Arms: 8X level

SUMMARY:
Exosomes are naturally occurring nanosized vesicles and comprised of natural lipid bilayers with the abundance of adhesive proteins that readily interact with cellular membranes. These vesicles have a content that includes cytokines and growth factors, signaling lipids, mRNAs, and regulatory miRNAs. Exosomes are involved in cell-to-cell communication, cell signaling, and altering cell or tissue metabolism at short or long distances in the body, and can influence tissue responses to injury, infection, and disease.

Experimental studies have demonstrated that mesenchymal stem cells (MSCs) or their exosomes (MSCs-Exo) significantly reduced lung inflammation and pathological impairment resulting from different types of lung injury. In addition, macrophage phagocytosis, bacterial killing and outcome were improved. It is highly likely that MSCs-Exo have the similar therapeutic effect on inoculation pneumonia as MSCs themselves.

This clinical study will be performed to evaluate the safety and tolerance of aerosol inhalation of the exosomes derived from allogenic adipose mesenchymal stem cells (MSCs-Exo) in healthy volunteers.

DETAILED DESCRIPTION:
Experimental studies have demonstrated that mesenchymal stem cells (MSCs) or their exosomes (MSCs-Exo) significantly reduced lung inflammation and pathological impairment resulting from different types of lung injury. In addition, macrophage phagocytosis, bacterial killing and outcome were improved. It is highly likely that MSCs-Exo have the similar therapeutic effect on inoculation pneumonia as MSCs themselves.

Although human bone marrow MSCs have been safely administered in patients with ARDS and septic shock (phase I/II trials), it seems safer to deliver MSCs-Exo rather than live MSCs. The intravenous administration of MSCs may result in aggregating or clumping in the injured microcirculation and carries the risk of mutagenicity and oncogenicity, which do not exist by treating with nebulized MSCs-Exo. Another advantage of MSCs-Exo over MSCs is the possibility of storing them for several weeks/months allowing their safe transportation and delayed therapeutic use.

The purpose of this study, therefore, is to explore the safety and efficiency as well as provide a clinical dose reference for the subsequent trails of aerosol inhalation of MSCs-Exo in the treatment of severe lung diseases (including severe lung infection, acute respiratory distress syndrome (ARDS) and chronic obstructive pulmonary disease (COPD), etc.)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers.
2. Age: 19-45, males and females.
3. The weight is within ± 10% of the standard weight [standard weight (kg) = 0.7 × (height cm-80)].
4. Examination indices of heart, liver, kidney and blood are all within the normal range.
5. According to Good Clinical Practice (GCP), volunteers who understand and voluntarily sign the consent form before this study.

Exclusion Criteria:

1. Women in pregnancy or lactation.
2. Primary diseases of important organs.
3. Mentally or physically disabled patients.
4. Suspected or definite history of alcohol and drug abuse.
5. According to the investigator's judgment, there is a low possibility of enrollment (such as frailty, etc.).
6. Volunteers who are allergic to the components of this medicine, or have a history of allergies to two or more drugs or food.
7. Volunteers who have diseases (such as insomnia) and are using other preventive and therapeutic drugs before this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jieming Qu, MD,PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Shi MM, Yang QY, Monsel A, Yan JY, Dai CX, Zhao JY, Shi GC, Zhou M, Zhu XM, Li SK, Li P, Wang J, Li M, Lei JG, Xu D, Zhu YG, Qu JM. Preclinical efficacy and clinical safety of clinical-grade nebulized allogenic adipose mesenchymal stromal cells-derived extracellular vesicles. J Extracell Vesicles. 2021 Aug;10(10):e12134. doi: 10.1002/jev2.12134. Epub 2021 Aug 14. PMID 34429860

RESULTS

PARTICIPANT FLOW:
Groups:
- 1X Level: Aerosol inhalation of MSCs-derived exosomes treatment participants will receive once aerosol inhalation of MSCs-derived exosomes (2.0*10E8 nano vesicles/3 ml)
  1X level of MSCs-Exo: Once aerosol inhalation of MSCs-derived exosomes (2.0*10E8 nano vesicles/3 ml)
- 2X Level: Aerosol inhalation of MSCs-derived exosomes treatment participants will receive once aerosol inhalation of MSCs-derived exosomes (4.0*10E8 nano vesicles/3 ml)
  2X level of MSCs-Exo: Once aerosol inhalation of MSCs-derived exosomes (4.0*10E8 nano vesicles/3 ml)
- 4X Level: Aerosol inhalation of MSCs-derived exosomes treatment participants will receive once aerosol inhalation of MSCs-derived exosomes (8.0*10E8 nano vesicles/3 ml)
  4X level of MSCs-Exo: Once aerosol inhalation of MSCs-derived exosomes (8.0*10E8 nano vesicles/3 ml)
- 6X Level: Aerosol inhalation of MSCs-derived exosomes treatment participants will receive once aerosol inhalation of MSCs-derived exosomes (12.0*10E8 nano vesicles/3 ml)
  6X level of MSCs-Exo: Once aerosol inhalation of MSCs-derived exosomes (12.0*10E8 nano vesicles/3 ml)
- 8X Level: Aerosol inhalation of MSCs-derived exosomes treatment participants will receive once aerosol inhalation of MSCs-derived exosomes (16.0*10E8 nano vesicles/3 ml)
  8X level of MSCs-Exo: Once aerosol inhalation of MSCs-derived exosomes (16.0*10E8 nano vesicles/3 ml)
Period: Overall Study
Arm/Group | 1X Level | 2X Level | 4X Level | 6X Level | 8X Level
Started | 3 | 3 | 6 | 6 | 6
Completed | 3 | 3 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1X Level | 2X Level | 4X Level | 6X Level | 8X Level | Total
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 24
Age, Continuous [Median (Full Range); unit: years] | 26 [25 to 34] | 26 [24 to 27] | 25 [21 to 35] | 25 [24 to 29] | 25.5 [24 to 27] | 25 [21 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 3 | 3 | 11
  Male | 1 | 2 | 4 | 3 | 3 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 3 | 3 | 6 | 6 | 6 | 24
Region of Enrollment [Number; unit: participants]
  China | 3 | 3 | 6 | 6 | 6 | 24
Comorbidity [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0 | 0 | 0
Smoking history [Count of Participants; unit: Participants] | 0 | 0 | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Reaction (AE) and Severe Adverse Reaction (SAE)
Description: Safety evaluation within 7 days after first treatment, including frequency of adverse reaction (AE) and severe adverse reaction (SAE)
Time Frame: from Day 0 to Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | 1X Level | 2X Level | 4X Level | 6X Level | 8X Level
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6
Participants | 1 | 0 | 0 | 0 | 1

2. Other Pre Specified Outcome: Alanine Aminotransferase (ALT) (IU/L)
Description: one of the indexes about liver function
Time Frame: day 0 and day 7
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | 1X Level | 2X Level | 4X Level | 6X Level | 8X Level
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6
IU/L
  Day 0 | 16 [16 to 24] | 21 [8 to 30] | 24 [14.25 to 42] | 17.5 [9.75 to 21.25] | 15.5 [13.25 to 18.5]
  Day 7 | 20 [16 to 21] | 24 [9 to 24] | 23.5 [13.25 to 58.25] | 16 [11.75 to 23.75] | 15.5 [11 to 18]

3. Other Pre Specified Outcome: Creatinine (Cr) (μmol/L)
Description: One of the indexes about kidney function
Time Frame: day 0 and day 7
Measure: Median (Inter-Quartile Range); unit: μmol/L
Arm/Group | 1X Level | 2X Level | 4X Level | 6X Level | 8X Level
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6
μmol/L
  Day 0 | 67 [64 to 86] | 83 [57 to 106] | 82.5 [62.75 to 90] | 74.5 [59 to 95] | 81 [56 to 91]
  Day 7 | 64 [59 to 86] | 77 [67 to 115] | 86 [63.25 to 92.75] | 74.5 [64.75 to 86.25] | 80 [56.5 to 90]

ADVERSE EVENTS:
Time Frame: 7days
Arm/Group | 1X Level | 2X Level | 4X Level | 6X Level | 8X Level
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/6 | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1X Level (N=3) | 2X Level (N=3) | 4X Level (N=6) | 6X Level (N=6) | 8X Level (N=6)
Sinus bradycardia (Cardiac disorders) | 1 (1) | NA | NA | NA | 1 (1) — Two subjects developed sinus bradycardia (58bpm, 59bpm) on the seventh day after nebulization according to EKG: one is in 1X group; the other is in 8X group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT04313647/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT04313647/ICF_001.pdf